CLINICAL TRIAL: NCT02507479
Title: Phase II Trial of Fludarabine Combined With Intravenous Thiotepa and Allogeneic Hematopoietic Stem-cell Transplantation in Patients With Lymphatic Malignancies Including Multiple Myeloma, Non Hodgkin's, Hodgkin Lymphoma and CLL
Brief Title: Thiotepa-based Conditioning for Allogeneic Stem-cell Transplantation (SCT) in Lymphoid Malignancies
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-13-0874-AN-CTIL
Record Dates: First submitted 2015-06-14; First posted 2015-07-24 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Non Hodgkin Lymphoma; Hodgkin Lymphoma; Chronic Lymphocytic Leukemia; Multiple Myeloma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma | interventions — Thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- thiotepa (Experimental): Thiotepa 5-10 mg/kg/d x 2 days
  Interventions: Drug: Thiotepa

INTERVENTIONS:
Drug: Thiotepa — Chemotherapy given prior to allogeneic stem cell transplantation

SUMMARY:
The study hypotheses is that the introduction of dose escalated thiotepa, in substitution to busulfan or melphalan, will reduce toxicity after allogeneic transplantation while improving disease eradication in patients with lymphoid malignancies not eligible for standard transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Age less than physiologic 68 years.
2. Patients with MM, NHL, HL and CLL with an indication for allogeneic transplantation as follows:

   1. MM; patients relapsing after autologous transplant or with high-risk cytogenetic abnormalities
   2. Aggressive lymphoma and Hodgkin lymphoma; relapse after autologous transplants
   3. Follicular lymphoma; failure of at least one prior regimen
   4. CLL; failure of prior therapy which includes Fludarabine combinations or 17p- cytogenetic abnormality
3. Patients must have an HLA matched related or unrelated donor willing to donate either peripheral blood stem cells or bone marrow. Matching is based on high-resolution class I (HLA-A, -B, -C) and class II (HLA-DRB1, -DQB) typing. The goal is to transplant > 3 x 106 CD34+ cells per kg body weight of the recipient
4. Patients must sign written informed consent.
5. Adequate birth control in fertile patients.

Exclusion Criteria:

1. Bilirubin > 3.0 mg/dl, transaminases > 3 times upper normal limit
2. Creatinine > 2.0 mg/dl
3. ECOG-Performance status > 2
4. Uncontrolled infection
5. Pregnancy or lactation
6. Abnormal lung diffusion capacity (DLCO < 40% predicted)
7. Severe cardiovascular disease
8. CNS disease involvement
9. Pleural effusion or ascites > 1 liter
10. Known hypersensitivity to Fludarabine or treosulfan
11. Psychiatric conditions/disease that impair the ability to give informed consent or to adequately co-operate

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 2 years after transplantation
  The percentage of patients alive without disease recurrence 2 years after transplant

SECONDARY OUTCOMES:
treatment-related mortality | 2 years after transplantation
  The percentage of patients who die of complications related to the transplant
graft versus host disease | 1 year after transplantation
  The percentage of patients experiencing graft-versus-host disease after transplant
relapse | 2 years after transplantation
  The percentage of patients experiencing disease recurrence after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Nagler, MD, Principal Investigator — Chaim Sheba Medical Center
Locations (1):
- Chaim Sheba Medical Center, Tel Litwinsky, Israel